CLINICAL TRIAL: NCT03653702
Title: Radiation-Free Technique for Evaluating Renal Scarring (RAFTERS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Richard Lee, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P00027566
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Vesico-Ureteral Reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contrast Enhanced Ultrasound (Experimental): Participants will undergo a contrast enhanced ultrasound (CEUS) using Lumason
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — Lumason will be used as the contrast agent. Standard Lumason dose will be used: 0.03mL/kg up to a maximum dose of 2.4 milliliter (mL) per injection

SUMMARY:
In this research study the investigators want to study a safe, radiation-free technique known as contrast-enhanced ultrasound that may improve the ability to diagnose or evaluate renal scarring compared to regular ultrasound. This technique requires injection into a vein of a small amount of contrast material called Lumason. Contrast material is a type of dye that helps the investigators image the structures in the body more clearly. If this technique is successful, the need for DMSA studies may be avoided to diagnose or evaluate kidney scarring. DMSA is a more expensive test, causes radiation exposure, may require sedation and/or injection of contrast agents with the potential to cause allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* patients older than or equal to 6 months and less than or equal to 35 years old and scheduled for Boston Children's Hospital (BCH) DMSA scan to evaluate renal function and/or renal scarring

Exclusion Criteria:

* patients with significant congenital renal anatomical abnormalities including horseshoe kidney, kidney malrotation, and multicystic dysplastic kidney (MCDK). Patients with severe cardio-pulmonary diseases will also be excluded.

Ages: 6 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Performance of CEUS result and comparison to DMSA | 3 months after final participant completes participation
  DMSA will be used as gold standard to evaluate CEUS test performance. Sensitivity and specificity of CEUS renal scarring detection will be calculated accordingly. Bivariate and multivariate analyses will be completed to compare patient characteristics between those with good and poor CEUS performance to investigate if CEUS performs better in patients with specific covariates

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States